CLINICAL TRIAL: NCT04396756
Title: A Randomized, Double-blind, Dose-ranging, Placebo Controlled Phase 2a Evaluation of the Safety, Tolerability and Pharmacokinetics of PLN-74809 in Participants With Idiopathic Pulmonary Fibrosis (INTEGRIS-IPF)
Brief Title: Evaluation of Efficacy and Safety of PLN-74809 in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLN-74809-IPF-202; INTEGRIS-IPF (Other: Pliant Therapeutics)
Record Dates: First submitted 2020-05-06; First posted 2020-05-21 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo
- PLN-74809 Dose Level 1 (Part A) (Experimental): PLN-74809 Dose Level 1 (Part A) - 4 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 Dose Level 2 (Part A) (Experimental): PLN-74809 Dose Level 2 (Part A) - 4 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 Dose Level 2 (Part B) (Experimental): PLN-74809 Dose Level 2 (Part B) - 12 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 - Dose Level 3 (Part C) (Experimental): PLN-74809 Dose Level 3 (Part C) - 12 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 - Dose Level 4 (Part C) (Experimental): PLN-74809 Dose Level 4 (Part C) - 12 weeks
  Interventions: Drug: PLN-74809
- PLN-74809 - Dose Level 5 (Part D) (Experimental): PLN-74809 Dose Level 5 (Part D) - ≥ 24 weeks
  Interventions: Drug: PLN-74809

INTERVENTIONS:
Drug: PLN-74809 — PLN-74809
  Arms: PLN-74809 - Dose Level 3 (Part C); PLN-74809 - Dose Level 4 (Part C); PLN-74809 - Dose Level 5 (Part D); PLN-74809 Dose Level 1 (Part A); PLN-74809 Dose Level 2 (Part A); PLN-74809 Dose Level 2 (Part B)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 2a, multicenter, 4-part, randomized, double-blind, dose-ranging, placebo-controlled study to evaluate the safety, tolerability, and PK of once-daily treatment with PLN-74809 in participants with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
Four part study:

Part A - 4 week treatment period evaluating PLN-74809 or matching placebo

Part B - 12 week treatment period evaluating PLN-74809 or matching placebo

Part C - 12 week treatment period evaluating up to two intermediatery PLN-74809 doses or matching placebo

Part D - ≥ 24 week treatment period evaluating higher PLN-74809 dose or matching placebo

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF based upon the Fleischner Society guidelines within 3 years from Screening (Part A) or based on ATS/ERS/JRS/ALAT 2018 guidelines within 5 years from Screening (Part B, C & D)
* FVC % of predicted ≥45%
* DLco (hemoglobin-adjusted) ≥30%
* Participants receiving treatment for IPF with nintedanib or pirfenidone are allowed, if on a stable dose for at least 3 months

Exclusion Criteria:

* Currently receiving or planning to initiate treatment for IPF (fibrosis) with agents not approved for that indication by the FDA
* Forced expiratory volume during the first seconds of the forced breath (FEV1)/FVC ratio <0.7 at Screening
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis that can affect FVC measurement or IPF progression
* Known acute IPF exacerbation or suspicion by the Investigator of such, within 6 months of Screening
* Smoking of any kind within 3 months of Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics Medical Monitor, Study Director — Pliant Therapeutics, Inc.
Locations (20):
- United States (10):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Interstitial Lung Disease Program, Pulmonary and Critical Care Medicine, Los Angeles, California
  - Yale University Scool of Medicine/ Yale New Haven Hospital, New Haven, Connecticut
  - The Emory Clinic, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cardio-Pulmonary Associates of St. Luke's Hospital - Chesterfield, Chesterfield, Missouri
  - PulmonIx, Greensboro, North Carolina
  - UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Lung Institute at One Hundred Oaks, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Dr. Anil Dhar Medicine Professional Corporation, Windsor, Ontario
  - CISSS de la Montérégie Centre, Greenfield Park, Quebec
- San Giuseppe Hospital, Multimedica S.p.a., Milan, Italy
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven, EJ
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, SZ
- New Zealand (2):
  - New Zealand Respiratory and Sleep Institute, Greenlane, Auckland
  - University of Otago Christchurch, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lancaster L, Cottin V, Ramaswamy M, Wuyts WA, Jenkins RG, Scholand MB, Kreuter M, Valenzuela C, Ryerson CJ, Goldin J, Kim GHJ, Jurek M, Decaris M, Clark A, Turner S, Barnes CN, Achneck HE, Cosgrove GP, Lefebvre EA, Flaherty KR; PLN-74809-IPF-202 Trial Investigators. Bexotegrast in Patients with Idiopathic Pulmonary Fibrosis: The INTEGRIS-IPF Clinical Trial. Am J Respir Crit Care Med. 2024 Aug 15;210(4):424-434. doi: 10.1164/rccm.202403-0636OC. PMID 38843105

RESULTS

PARTICIPANT FLOW:
Groups:
- PLN-74809 (Part A) - 40 mg: PLN-74809 (Part A): Consists of an up to 28-day screening period, a 4-week treatment period, and a 2-week (+/- 3 days) post-treatment follow-up period.
  PLN-74809 tablet administered orally.
  Participants took either PLN-74809 40mg or a matching placebo with 100ml water after fasting.
- PLN-74809 (Part B) - 40 mg: PLN-74809 (Part B): Consists of an up to 28-day screening period, a 12-week treatment period, and a 2-week (+/- 3 days) post-treatment follow-up period.
  PLN-74809 tablet administered orally.
  Participants took either PLN-74809 40mg or a matching placebo with 240ml water after fasting.
- PLN-74809 (Part C) - 80 mg: PLN-74809 (Part C): Consists of an up to 28-day screening period, a 12-week treatment period, and a 2-week (+/- 3 days) post-treatment follow-up period.
  PLN-74809 tablet administered orally.
  Participants took either PLN-74809 80mg or a matching placebo with 240ml water after fasting.
- PLN-74809 (Part C) - 160 mg: PLN-74809 (Part C): Consists of an up to 28-day screening period, a 12-week treatment period, and a 2-week (+/- 3 days) post-treatment follow-up period.
  PLN-74809 tablets administered orally.
  Participants took either PLN-74809 160mg or a matching placebo with 240ml water after fasting.
- PLN-74809 (Part D) -320 mg: PLN-74809 (Part D): Consists of an up to 28-day screening period, at least 24-week treatment period, and a 2-week (+/- 3 days) post-treatment follow-up period.
  PLN-74809 tablets administered orally.
  Participants took either PLN-74809 320 mg or a matching placebo with 240ml water after fasting.
- Placebo: Matching placebo tablets administered orally.
  Participants took a matching placebo with water after fasting.
Period: Overall Study
Arm/Group | PLN-74809 (Part A) - 40 mg | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) -320 mg | Placebo
Started | 1 | 22 | 23 | 22 | 21 | 31
Received Placebo | 0 | 0 | 0 | 0 | 1 | 0
Completed | 1 | 21 | 23 | 20 | 15 | 25
Not Completed | 0 | 1 | 0 | 2 | 6 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who took at least 1 dose of study drug.
  Overall Number of Participants is 120 not 121. One participant received both placebo and PLN-74809 320 mg due to incorrect study drug dispensation and is counted in the denominator of both treatment groups for demographic and safety reporting.
Groups:
- PLN-74809 (Part A) - 40 mg: PLN-74809 (Part A) - 40 mg PLN-74809
- PLN-74809 (Part B) - 40 mg: PLN-74809 (Part B) - 40 mg PLN-74809
- PLN-74809 (Part C) - 80 mg: PLN-74809 (Part C) - 80 mg PLN-74809
- PLN-74809 (Part C) - 160 mg: PLN-74809 (Part C) - 160 mg PLN-74809
- PLN-74809 (Part D) - 320 mg: PLN-74809 (Part D) - 320 mg PLN-74809
- Placebo: Placebo (Part B, C, D)
- Total: Total of all reporting groups
Arm/Group | PLN-74809 (Part A) - 40 mg | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) - 320 mg | Placebo | Total
Number analyzed (Participants) | 1 | 22 | 23 | 22 | 21 | 31 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (NA) — No SD due to only 1 data point available | 69.2 (7.11) | 74.2 (4.70) | 71.5 (6.63) | 70.6 (7.31) | 72.1 (6.20) | 71.4 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 6 | 1 | 4 | 19
  Male | 1 | 18 | 19 | 16 | 20 | 27 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 21 | 23 | 22 | 21 | 31 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 22 | 21 | 22 | 20 | 30 | 116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A - Number of Participants With Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant administered a study drug that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not the AE is considered related to the study drug. TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 14 days after permanent discontinuation of study drug.
Time Frame: Up to 4 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- PLN-74809 (Part A) - 40 mg: PLN-74809 (Part A) - up to 4 weeks
  40 mg PLN-74809
Arm/Group | PLN-74809 (Part A) - 40 mg
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Part B, C, D - Number of Participants With Treatment-Emergent Adverse Events
Description: as for outcome 1
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- PLN-74809 (Part B) - 40 mg: PLN-74809 (Part B) - up to 12 weeks
  40 mg PLN-74809
- PLN-74809 (Part C) - 80 mg: PLN-74809 (Part C) - up to 12 weeks
  80 mg PLN-74809
- PLN-74809 (Part C) - 160 mg: PLN-74809 (Part C) - up to 12 weeks
  160 mg PLN-74809
- PLN-74809 (Part D) - 320 mg: PLN-74809 (Part D) - at least 24 weeks and up to 48 weeks
  320 mg PLN-74809
- Placebo (Part B, C, D): Placebo (Part B, C) - up to 12 weeks
  Placebo (Part D) - at least 24 weeks and up to 48 weeks
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) - 320 mg | Placebo (Part B, C, D)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 31
Participants | 16 | 15 | 14 | 17 | 21

3. Primary Outcome: Part D - Number of Participants With Treatment-Emergent Adverse Events
Description: as for outcome 1
Time Frame: Up to 48 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- PLN-74809 (Part D) -320 mg: PLN-74809 (Part D) - at least 24 weeks and up to 48 weeks
  320 mg PLN-74809
- Placebo (Part D): Placebo (Part D) - at least 24 weeks and up to 48 weeks
Arm/Group | PLN-74809 (Part D) -320 mg | Placebo (Part D)
Number analyzed (Participants) | 22 | 8
Participants | 20 | 7

4. Primary Outcome: Part A - Number of Participants With Serious Treatment-Emergent Adverse Events
Description: An SAE was defined as an event that, at any dose, results in the following: death, a life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect or a medically important event or reaction.
Time Frame: Up to 4 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PLN-74809 (Part A) - 40 mg
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Part B, C, D - Number of Participants With Serious Treatment-Emergent Adverse Events
Description: as for outcome 4
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) -320 mg | Placebo (Part B, C, D)
Number analyzed (Participants) | 22 | 23 | 22 | 22 | 31
Participants | 1 | 0 | 2 | 1 | 3

6. Primary Outcome: Part D - Number of Participants With Serious Treatment-Emergent Adverse Events
Description: as for outcome 4
Time Frame: Up to 48 weeks
Population: Safety Population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PLN-74809 (Part D) -320 mg | Placebo (Part D)
Number analyzed (Participants) | 22 | 8
Participants | 2 | 1

7. Secondary Outcome: Part A - Assessment of PLN-74809 Total Plasma Concentrations
Description: Part A - Assessment of PLN-74809 Total Plasma Concentrations Week 4, 1 Hour Post Dose
Time Frame: Week 4, 1 Hour Post Dose
Population: Pharmacokinetic Population included all participants who took at least 1 dose of study drug with at least one post baseline evaluable PLN-74809 concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLN-74809 (Part A) - 40 mg
Number analyzed (Participants) | 1
ng/mL | 829 (NA) — SD is NA due to only 1 data point available

8. Secondary Outcome: Part B, C, D - Assessment of PLN-74809 Total Plasma Concentrations
Description: Part B, C, D - Assessment of PLN-74809 Total Plasma Concentrations Week 12, 2 Hours Post Dose
Time Frame: Week 12, 2 Hours Post Dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) - 320 mg
Number analyzed (Participants) | 20 | 23 | 21 | 18
ng/mL | 921.45 (549.103) | 1731.70 (875.776) | 2733.71 (1038.402) | 3742.78 (1383.345)

9. Secondary Outcome: Part D - Assessment of PLN-74809 Total Plasma Concentrations
Description: Part D - Assessment of PLN-74809 Total Plasma Concentrations Week 24, 2 Hours Post Dose
Time Frame: Week 24, 2 Hours Post Dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLN-74809 (Part D) - 320 mg
Number analyzed (Participants) | 16
ng/mL | 4120.63 (1866.606)

10. Other Pre Specified Outcome: Part B, C, D - Assessment of Change From Baseline in Forced Vital Capacity (FVC)
Description: Change from Baseline by Visit, Mixed Model for Repeated Measures through Week 12.
Time Frame: Up to 12 weeks
Population: Efficacy modified Intent-to-Treat (mITT) Population includes all randomized participants who do not have FVC values that meet outlier criteria.
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- PLN-74809 (Part D) -320 mg: PLN - 74809 (Part D) - at least 24 weeks and up to 48 weeks
  320 mg PLN-74809
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) -320 mg | Placebo (Part B, C, D)
Number analyzed (Participants) | 21 | 23 | 21 | 18 | 25
mL | -46.1 (39.64) | 25.6 (38.57) | -25.6 (40.49) | 29.4 (43.35) | -110.5 (36.38)

11. Other Pre Specified Outcome: Part D - Assessment of Change From Baseline in Forced Vital Capacity (FVC)
Description: Change from Baseline by Visit, Mixed Model for Repeated Measures through Week 24.
Time Frame: Up to 24 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | PLN-74809 (Part D) -320 mg | Placebo (Part D)
Number analyzed (Participants) | 16 | 6
mL | -35.9 (50.57) | -109.3 (74.93)

12. Other Pre Specified Outcome: Part B, C, D - Change in Pulmonary Fibrosis Score by Quantitative HRCT at Week 12
Description: Quantitative Lung Fibrosis extent (%) measures the percentage of lung tissue that is assessed as fibrotic.
Time Frame: Up to 12 weeks
Population: Per computed tomography (CT) population includes all randomized participants with evaluable CT scans per the imaging charter.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) - 320 mg | Placebo (Part B, C, D)
Number analyzed (Participants) | 15 | 18 | 14 | 16 | 25
Percentage | 3.15 (4.796) | 0.70 (4.194) | 0.00 (3.960) | 0.20 (2.817) | 1.46 (4.951)

13. Other Pre Specified Outcome: Part D - Change in Pulmonary Fibrosis Score by Quantitative HRCT at Week 24
Description: Quantitative Lung Fibrosis extent (%) measures the percentage of lung tissue that is assessed as fibrotic.
Time Frame: Up to 24 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | PLN-74809 (Part D) -320 mg | Placebo (Part D)
Number analyzed (Participants) | 14 | 6
Percentage | 1.31 (2.650) | 3.72 (4.381)

14. Other Pre Specified Outcome: Part B,C, D - Assessment of Change From Baseline in a Visual Analog Scale (VAS) Scale for Cough
Description: Visual Analog Scale for Cough measures participant reported cough severity on a scale of 0 to 100 with higher scores representative of more severe cough. A negative change from baseline nominally represents reduced cough severity and a positive change from baseline nominally represents increased cough severity.
Time Frame: Up to 12 weeks
Population: Efficacy Intent-to-Treat (ITT) Population includes all randomized participants with evaluable cough scores.
Measure: Mean (Standard Deviation); unit: Point
Arm/Group | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) - 160 mg | PLN-74809 (Part D) - 320 mg | Placebo (Part B, C, D)
Number analyzed (Participants) | 21 | 23 | 21 | 18 | 28
Point | 1.2 (20.92) | 0.7 (13.85) | 3.8 (26.46) | -2.9 (31.19) | -0.3 (16.43)

15. Other Pre Specified Outcome: Part D - Assessment of Change From Baseline in a Visual Analog Scale (VAS) Scale for Cough
Description: as for outcome 14
Time Frame: Up to 24 weeks
Population: Efficacy Intent-to-Treat (ITT) Population includes all randomized participants with evaluable cough scores.
Measure: Mean (Standard Deviation); unit: Point
Arm/Group | PLN-74809 (Part D) -320 mg | Placebo (Part D)
Number analyzed (Participants) | 16 | 5
Point | -1.9 (17.70) | 16.8 (33.78)

ADVERSE EVENTS:
Time Frame: All cause mortality: randomization up to 190.1 days plus 14 days. Adverse events: First dose date up to 29 days plus 14 days (Part A PLN-74809 40 mg), up to 83.6 days plus 14 days (Part B PLN-74809 40 mg), up to 86.0 days plus 14 days (Part C PLN-74809 80 mg), up to 82.7 days plus 14 days (Part C PLN-74809 160 mg), up to 190.1 days plus 14 days (Part D PLN-74809 320 mg) and up to 107.6 days plus 14 days (Parts B, C, D placebo).
Description: All-cause mortality: All Randomized population included all participants who were randomized in the study.
  Adverse Events: Safety population included all participants who took at least 1 dose of study drug.
Groups:
- PLN-74809 (Part C) -160 mg: PLN-74809 (Part C) -160 mg PLN-74809
Arm/Group | PLN-74809 (Part A) - 40 mg | PLN-74809 (Part B) - 40 mg | PLN-74809 (Part C) - 80 mg | PLN-74809 (Part C) -160 mg | PLN-74809 (Part D) - 320 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/22 | 0/23 | 0/22 | 1/22 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/22 | 0/23 | 2/22 | 2/22 | 3/31
Other Adverse Events (participants affected / at risk) | 1/1 | 8/22 | 8/23 | 10/22 | 18/22 | 14/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLN-74809 (Part A) - 40 mg (N=1) | PLN-74809 (Part B) - 40 mg (N=22) | PLN-74809 (Part C) - 80 mg (N=23) | PLN-74809 (Part C) -160 mg (N=22) | PLN-74809 (Part D) - 320 mg (N=22) | Placebo (N=31)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis/Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLN-74809 (Part A) - 40 mg (N=1) | PLN-74809 (Part B) - 40 mg (N=22) | PLN-74809 (Part C) - 80 mg (N=23) | PLN-74809 (Part C) -160 mg (N=22) | PLN-74809 (Part D) - 320 mg (N=22) | Placebo (N=31)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 5 (8) | 7 (11) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 3 (3)
Idiopathic pulmonary fibrosis/Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 4 (4) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, the data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Any publication of the results of this study must be authorized by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04396756/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04396756/SAP_001.pdf